CLINICAL TRIAL: NCT01870414
Title: Electromyographic Analysis And Body Balance In The Use Of Athletes After Cryotherapy By Immersion Ankle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1143-6567
Record Dates: First submitted 2013-05-28; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Individual Adjustment; Itch; Athlete
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cryotherapy by immersion (Other): the dominant leg was immersed in cold water for 20 minutes [2, 17], temperature of 4º C [22, 24], water level at 20 cm.
  Interventions: Other: cryotherapy by immersion

INTERVENTIONS:
Other: cryotherapy by immersion — the dominant leg was immersed in cold water for 20 minutes [2, 17], temperature of 4º C [22, 24], water level at 20 cm
  Other Names: Cryoimmersion, 20 minutes, temperature was 4C.

SUMMARY:
The influence of cryotherapy on ankle motor control and balance of athletes is controversial. The aim of this study is to assess the neuromuscular response of the dominant leg and body balance basketball athletes after application of cryotherapy. The sample is distributed into two groups. Group one will consist of 20 basketball players without a history of ankle sprains in the past 12 months and no complaints of instability in this joint, and group two, 20 non-athletes, active, no complaints in the lower limb in the last 12 months. Will perform the inversion movements and single-leg hop for the analysis of the electromyographic signal of anterior tibial, peroneal, gastrocnemius (lateral), rectus femoris, hamstrings and gluteus medius. Will also be performed kinematic analysis in search of body balance and range of motion of the joints of the lower limbs. And yet, the analysis of the plantar support and ground reaction force. After the initial collection of the data subjects will be submitted to the application of cryotherapy by immersion in a time of 20 minutes, with a temperature of 6 ± 2 degrees Celsius. Data collection will be held in pre, 0, 10, 20 and 30 minutes after application of cryotherapy. The data will be statistically analyzed to compare the results in collection times within and between groups. The significance level is set at 5%. The data support the intended use of cryotherapy in motor control of the inversion movement, jump and balance of athletes.

DETAILED DESCRIPTION:
Forty male subjects, aged 21.6 (±3.2) yr, 177.9 (±7.9) cm tall, 82.8 (±19.3) Kg body weight and 25.9 (±4.8) Kg.m-2 body mass index (BMI) were evaluated. Skin surface temperature before and after cold-water immersion was 27.7(±3)°C and 7.1 (±1)°C, respectively (p=0,0001).

ELIGIBILITY:
Inclusion Criteria:Healthy, active individuals and athletes basketball. -

Exclusion Criteria:patients with muscle or joint injuries in the lower limbs in the last six months; metabolic diseases, rheumatic and orthopedic disabling; patients with balance disorders or cognitive; individuals to submit complaints of muscle fatigue at the time of the tests or they needed the use of stabilizers to realize them; subjects with skin lesions of the lower extremities, hypersensitivity to cold and suffering from Diabetes Mellitus.

-

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Cryoimmersion decreases neuromuscular response of lower limb after ankle inversion | 2 years
  The peak values of the electromyographic signal amplitude (RMS) were obtained from thirty-five healthy, active university subjects after the use of a tilt platform to force the ankle into a 30º of inversion before (pre), and immediately after (post) 10, 20, and 30 minutes, followed by cold-water immersion at 4ºC, for 20 minutes. Shapiro-Wilk test, Repeated Measure Analysis and Bonferroni post-hoc test provided the results. Peak RMS values were significantly lower at all times after cold-water immersion when compared to prior application for all muscles, except in the post-immediate time for GM. There was a decrease in muscular response to the ankle inversion movement after cooling, with residual effect of up to 30 minutes. Therefore, special care should be taken by those involved in sports activities.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Macedo, master, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Macedo CS, Alonso CS, Liporaci RF, Vieira F, Guirro RR. Cold water immersion of the ankle decreases neuromuscular response of lower limb after inversion movement. Braz J Phys Ther. 2014 Jan-Feb;18(1):93-7. doi: 10.1590/s1413-35552012005000132. Epub 2014 Jan 8. PMID 24675918